CLINICAL TRIAL: NCT02466373
Title: Pharmacokinetics and Clinical Effects of Escalating Doses of Clonidine in ICU Patients
Acronym: Clokin1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Deventer Ziekenhuis (Other)
Responsible Party: Principal Investigator, M. Zeeman, drs M. Zeeman, Deventer Ziekenhuis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clonidine kinetics 1.1
Record Dates: First submitted 2015-04-21; First posted 2015-06-09 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Delirium; Critical Illness
Keywords: clonidine; pharmacodynamics; pharmacokinetics; intensive care; delirium
MeSH Terms: conditions — Delirium; Critical Illness | interventions — Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- No clonidine (No Intervention): No clonidine is administered. The outcome measures are recorded, to compare them with the outcome measures of the other clonidine arms
- Clonidine 600mcg (Experimental): 4 patients receive 600 µg/day of clonidine without loading schedule. 4 patients receive 600 µg/day of clonidine with a loading schedule of 300 µg in 4 h.
  Interventions: Drug: Clonidine (Catapresan®) 0,150 mg/ml, ampoule 1 ml
- Clonidine 1200mcg (Experimental): * 4 patients receive 1200 µg/day of clonidine without loading schedule.
  * 4 patients receive 1200 µg/day of clonidine with a loading schedule of 600 µg in 4 h.
  Interventions: Drug: Clonidine (Catapresan®) 0,150 mg/ml, ampoule 1 ml
- Clonidine 1800mcg (Experimental): * 4 patients receive 1800 µg/day of clonidine without loading schedule.
  * 4 patients receive 1800 µg/day of clonidine with a loading schedule of 900 µg in 4 h.
  Interventions: Drug: Clonidine (Catapresan®) 0,150 mg/ml, ampoule 1 ml

INTERVENTIONS:
Drug: Clonidine (Catapresan®) 0,150 mg/ml, ampoule 1 ml — clonidine intravenous
  Other Names: Boehringer Ingelheim, RVG 06055
  Arms: Clonidine 1200mcg; Clonidine 1800mcg; Clonidine 600mcg

SUMMARY:
This study is developed for assessing the pharmacodynamic and pharmacokinetic properties of intravenous (IV) clonidine in critically ill patients on the ICU, and to estimate the optimal dosing strategy for IV clonidine.

DETAILED DESCRIPTION:
Many patients in intensive care units (ICU's) require sedation and analgesia to tolerate mechanical ventilation and other ICU procedures. Commonly used GABA-ergic anaesthetics like propofol, midazolam and morphine have potential adverse effects that may increase morbidity, prolong ICU stay and provoke delirium. Recent studies have shown that sedation with alpha-2-adrenergic agonists may lead to a reduction of the total amount of gamma-aminobutyric acid (GABA) -ergic anaesthetics and reduction of delirium1In clinical practice the alpha-2-adrenergic agent clonidine is widely used off label as an add-on sedative in mechanically ventilated patients who suffer from delirium, but there are no large studies proving that this therapy is effective and safe. Limited information exists on the pharmacokinetics of iv clonidine, especially in ICU patients. Besides, dosing regimens of clonidine differ widely among ICU's in the Netherlands, and in the literature.

The sample size required for pharmacokinetic modelling with an acceptable level of precision is inversely related to the number of blood samplings taken from each individual. Population pharmacokinetic experiments that have been published have generally used 50 or more subjects. However, in the investigators study a relatively large number of blood samples are taken (>10 per subject when the protocol is completed, see section 6.3). THe investigators estimate that sufficient precision can be obtained with a sample size of 24 subjects, generating an estimated 240 to 360 blood samples.

In a recent publication of a computer simulated population pharmacokinetics of an absorption model using a design that involved 6 samplings per subject, it was estimated that a two-compartment first-order model would need 50 subjects (i.e. 300 blood samplings) to obtain a model with 50% precision and a power of 0.8.

The investigators 24 subjects will be treated with 3 different doses of clonidine (600, 1200 and 1800 µg/day), that is 8 per treatment arm.

On top of this, 8 patients receiving no clonidine will serve as a reference group, in order to interpret hemodynamic and safety data, and to illustrate dose-response relationships.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must be:

* at least 18 years of age
* intubated
* sedated at the start of the study. Because of the high incidence of delirium on the ICU in all age categories, all age groups > 18 years will be included

Exclusion Criteria:

* Severe neurotrauma,
* Severe dementia (living in a nursing home)
* Inability to speak Dutch or English, which is one of the causes of not being able to use the CAM-ICU.
* The use of clonidine during the 96 hours before the start of the study.
* Bradycardia (<50/min)
* Severe hypotension (MAP < 65 after volume resuscitation and vasopressors)
* Pregnancy and lactation (pregnancy test are routinely performed in premenopausal women on the ICU).
* Epilepsy
* Known clonidine intolerance
* Liver cirrhosis (Child Pugh class C)
* Recent and acute myocardial infarction
* Severe heart failure (LVEF < 30%)
* Second or third degree atrioventricular (AV)-block without a permanent pacemaker
* Expected transfer to another hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-12; Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
clonidine plasma concentrations | up to 7 days
  pharmacokinetic and pharmacodynamic properties of intravenous clonidine in ICU patients Clonidine plasma concentration at start of infusion at t=2, t=4, t=8 and t=12 h Clonidine plasma concentration during study, once daily Clonidine plasma concentration after stopping infusion at t=ω+8, t=ω+16, t=ω+24 h, and t=ω+48 h (ω= end of infusion).

SECONDARY OUTCOMES:
heart rate | up to 7 days
  Heart rate 2-hrly for the first 12 h, 8-hrly thereafter
blood pressure | up to 7 days
  Blood pressure 2-hrly for the first 12 h, 8-hrly thereafter
delirium | up to 7 days
  delirium rating scale, CAM-ICU 3 times daily
use of antipsychotics | up to 7 days
  additional use of haloperidol or sedatives, measured in total amount during the investigational period

CONTACTS AND LOCATIONS:
Overall Officials: Huub Oever v/d, Principal Investigator — Deventer Ziekenhuis
Locations (1):
- Deventer Hospital, Deventer, Netherlands

IPD SHARING:
Plan to Share IPD: No